CLINICAL TRIAL: NCT01124838
Title: A Multicenter Study of the Efficacy and Safety of the Human Anti-TNF Monoclonal Antibody Adalimumab in Subjects With Inactive Non-infectious Intermediate Uveitis, Posterior Uveitis, or Panuveitis - Including a Sub-study in Japanese Patients
Brief Title: Efficacy and Safety of Adalimumab in Subjects With Inactive Uveitis
Acronym: Visual II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-880; 2009-016008-22 (EudraCT Number)
Record Dates: First submitted 2010-05-14; First posted 2010-05-17 (Estimated); Results first posted 2016-06-21 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Uveitis
Keywords: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Adalimumab; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection at Baseline followed by every other week (eow) dosing starting at Week 1 for up to 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 10 to 35 mg/day at study entry followed by a protocol-defined mandatory taper until Week 19.
  Interventions: Drug: Prednisone; Drug: Placebo
- Adalimumab (Experimental): Participants received adalimumab 80 mg subcutaneous loading dose at Baseline followed by 40 mg doses eow starting at Week 1 for a maximum of 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 10 - 35 mg/day at study entry followed by a protocol-defined mandatory taper until Week 19.
  Interventions: Drug: Adalimumab; Drug: Prednisone

INTERVENTIONS:
Drug: Adalimumab — Administered subcutaneously as an 80 mg loading dose (2 syringes) at Baseline followed by 40 mg eow starting at Week 1.
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab
Drug: Prednisone — Administered orally, 10 - 35 mg/day at study entry followed by a protocol-defined mandatory taper schedule in which all subjects continuing in the study were to discontinue prednisone no later than Week 19.
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
A study comparing the safety and efficacy of adalimumab compared with. placebo in adults with inactive non-infectious intermediate uveitis, posterior uveitis, or panuveitis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with non-infectious intermediate, posterior, or panuveitis.
* Subject that for ≥ 28 days prior to the Baseline visit has inactive disease and is taking ≥ 10 mg of oral prednisone to maintain this inactive state and fulfillment of all 3 of the following criteria based on the Investigator's clinical judgment at the Screening and Baseline visits for both eyes:

  * Subject without active, inflammatory chorioretinal and/or inflammatory retinal vascular lesions.
  * Subject with anterior chamber cell grade ≤ 0.5+ according to Standardization of Uveitis Nomenclature (SUN) criteria.
  * Subject with vitreous haze grade ≤ 0.5+ according to National Eye Institute (NEI)/SUN criteria.
* Subject is on oral prednisone 10 to 35 mg/day (or oral corticosteroid equivalent) at Baseline and the dose has not been increased in the past 28 days or decreased in the past 14 days.
* Subject must have a documented history of experiencing at least one disease flare within 18 months of the Screening visit. This flare has to occur during or up to a maximum of 28 days after tapering off the oral corticosteroid therapy.
* Subjects who do not have previous, active or latent tuberculosis (TB). Only one TB test is required to allow the subject in the study. Subjects with either negative purified protein derivative (PPD) (< 5 mm of induration) or negative QuantiFERON®-TB Gold test (or interferon-gamma release assay (IGRA) equivalent) are eligible. Subjects with a repeat indeterminate QuantiFERON®-TB Gold test (or IGRA equivalent) result are not eligible. Note, that only one TB screening test is allowed and required. A repeat QuantiFERON®-TB Gold test (or IGRA equivalent) is not permitted if the PPD skin test is positive. The TB screening tests are diagnostic tests. In the event of a negative TB screening test, the results are to be interpreted in the context of the patient's epidemiology, history, exam findings, etc. and it is the responsibility of the investigator to determine if a patient has previous, active or latent tuberculosis or not. Under no circumstances can a patient with a positive PPD result or positive QuantiFERON®-TB Gold test (or IGRA equivalent) enter the study.

Exclusion Criteria:

* Subject with isolated anterior uveitis.
* Subject with confirmed or suspected infectious uveitis, including but not limited to infectious uveitis due to TB, cytomegalovirus (CMV), Lyme disease, toxoplasmosis, human T-lymphotropic virus type 1 (HTLV-1) infection, Whipple's disease, herpes zoster virus (HZV) and herpes simplex virus (HSV).
* Subject with serpiginous choroidopathy.
* Subject with corneal or lens opacity that precludes visualization of the fundus or that likely requires cataract surgery during the duration of the trial.
* Subject with intraocular pressure of ≥ 25 mmHg and on ≥ 2 glaucoma medications or evidence of glaucomatous optic nerve injury.
* Subject with best corrected visual acuity (BCVA) less than 20 letters (ETDRS [Early Treatment Diabetic Retinopathy Study]) in at least one eye at the Baseline visit.
* Subject with intermediate uveitis or panuveitis that has signs of intermediate uveitis (e.g. presence or history of snowbanking or snowballs) and symptoms and/or magnetic resonance imaging (MRI) findings suggestive of a demyelinating disease such as multiple sclerosis. All subjects with intermediate uveitis or panuveitis that have signs of intermediate uveitis (e.g. presence or history of snowbanking or snowballs) must have a brain MRI within 90 days prior to the Baseline visit.
* Subject has previous exposure to anti-tumor necrosis factor (TNF) therapy or any biologic therapy (except intravitreal anti- vascular endothelial growth factor (VEGF) therapy) with a potential therapeutic impact on non-infectious uveitis.
* Subject on concomitant immunosuppressive therapy other than methotrexate, cyclosporine, mycophenolate mofetil or an equivalent drug to mycophenolate mofetil (e.g., mycophenolic acid), azathioprine or tacrolimus within 28 days of Baseline or has discontinued an immunosuppressive therapy including methotrexate, cyclosporine, mycophenolate mofetil or an equivalent drug to mycophenolate mofetil (e.g., mycophenolic acid), azathioprine or tacrolimus within 28 days of Baseline.
* If entering the study on one concomitant immunosuppressive therapy, dose has not been stable for at least 28 days prior to the Baseline visit or is not within the following allowable doses at the Baseline visit:

  * Methotrexate (MTX) ≤ 25 mg per week
  * Cyclosporine ≤ 4 mg/kg per day
  * Mycophenolate mofetil ≤ 2 grams per day or an equivalent drug to mycophenolate mofetil (e.g. mycophenolic acid) at an equivalent dose approved by the Medical Monitor
  * Azathioprine ≤ 175 mg per day
  * Tacrolimus (oral formulation) ≤ 8 mg per day
* Subject has Retisert® (glucocorticosteroids implant) within 3 years prior to the Baseline visit or has had complications related to the device. Subject has had Retisert® (glucocorticosteroid implant) removed within 90 days prior to the Baseline visit or has had complications related to removal of the device.
* Subject has received intraocular or periocular corticosteroids within 90 days prior to the Baseline visit.
* Subject with proliferative or severe non-proliferative diabetic retinopathy or clinically significant macular edema due to diabetic retinopathy.
* Subject with neovascular/wet age-related macular degeneration.
* Subject with abnormality of vitreo-retinal interface (i.e., vitreomacular traction, epiretinal membranes, etc.) with the potential for macular structural damage independent of the inflammatory process.
* Subject with cystoid macular edema unless the retinal changes are persistent, residual and stable as defined by the SUN criteria (persistent is > 3 months duration).
* Subject has received Ozurdex® (dexamethasone implant) within 6 months prior to the Baseline visit.
* Subject has received intravitreal methotrexate within 90 days prior to the Baseline visit.
* Subject has received intravitreal anti-VEGF therapy:

  * within 45 days of the Baseline visit for Lucentis® (ranibizumab) or Avastin® (bevacizumab);
  * or within 60 days of the Baseline visit for anti-VEGF Trap (Aflibercept).
* Subject on systemic carbonic anhydrase inhibitor within 1 week prior to Screening visit.
* Subject with a history of scleritis.
* Subject on cyclophosphamide within 30 days prior to the Baseline visit.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2010-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Payne, Study Director — AbbVie

REFERENCES:
- [Background] Nguyen QD, Merrill PT, Jaffe GJ, Dick AD, Kurup SK, Sheppard J, Schlaen A, Pavesio C, Cimino L, Van Calster J, Camez AA, Kwatra NV, Song AP, Kron M, Tari S, Brezin AP. Adalimumab for prevention of uveitic flare in patients with inactive non-infectious uveitis controlled by corticosteroids (VISUAL II): a multicentre, double-masked, randomised, placebo-controlled phase 3 trial. Lancet. 2016 Sep 17;388(10050):1183-92. doi: 10.1016/S0140-6736(16)31339-3. Epub 2016 Aug 16. PMID 27542302
- [Derived] Sheppard J, Joshi A, Betts KA, Hudgens S, Tari S, Chen N, Skup M, Dick AD. Effect of Adalimumab on Visual Functioning in Patients With Noninfectious Intermediate Uveitis, Posterior Uveitis, and Panuveitis in the VISUAL-1 and VISUAL-2 Trials. JAMA Ophthalmol. 2017 Jun 1;135(6):511-518. doi: 10.1001/jamaophthalmol.2017.0603. PMID 28426849
- See also: This clinical study may be evaluating a usage that is not currently FDA-approved. Please see US Prescribing Information for approved uses. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study includes a Japan sub-study. A total of 261 adults with inactive non-infectious intermediate uveitis, posterior uveitis or panuveitis were randomized at 72 study sites worldwide; 229 participants at 62 study sites in Australia, Israel, Latin America, North America, and Europe (Main Study), and 32 participants at 10 study sites in Japan.
Pre-assignment Details: Participants were randomized in a 1:1 ratio double-masked fashion using baseline immunosuppressant (IMM) usage as the stratification factor. Participants in the Japan sub-study were randomized in a separate stratum with no stratification by baseline IMM usage.
  Study completion is defined as meeting treatment failure or reaching study Week 80.
Period: Overall Study
Arm/Group | Placebo | Adalimumab
Started | 130 | 131
Enrolled in Main Study | 114 | 115
Enrolled in Japan Sub-study | 16 | 16
Completed | 112 | 116
Not Completed | 18 | 15
Not completed — Miscellaneous | 4 | 2
Not completed — Adverse Event | 7 | 11
Not completed — Lack of Efficacy | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab | Total
Number analyzed (Participants) | 130 | 131 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.22 (14.026) | 43.18 (12.719) | 43.20 (13.360)
Age, Customized [Number; unit: participants]
  < 65 years | 121 | 125 | 246
  ≥ 65 years | 9 | 6 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 75 | 158
  Male | 47 | 56 | 103
Race/Ethnicity, Customized [Number; unit: participants]
  White | 96 | 96 | 192
  Black | 8 | 6 | 14
  Asian | 19 | 19 | 38
  American Indian/Alaskan Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 5 | 9 | 14
  Multi-Race | 1 | 1 | 2
Type of Uveitis [Number; unit: participants]
  Intermediate | 30 | 17 | 47
  Posterior | 36 | 41 | 77
  Panuveitis | 63 | 71 | 134
  Intermediate/Posterior | 1 | 2 | 3
Diagnosis [Number; unit: participants]
  Idiopathic | 45 | 33 | 78
  Birdshot Choroidopathy | 16 | 15 | 31
  Multifocal Choroiditis and Panuveitis | 2 | 5 | 7
  Vogt Koyanagi Harada | 30 | 34 | 64
  Sarcoid | 20 | 22 | 42
  Behcet's | 7 | 10 | 17
  Other | 10 | 12 | 22
Eye Affected [Number; unit: participants]
  Left | 3 | 3 | 6
  Right | 5 | 2 | 7
  Both | 122 | 126 | 248
History of Infectious Uveitis [Number; unit: participants]
  Yes | 0 | 0 | 0
  No | 130 | 131 | 261
Duration of Uveitis [Mean (Standard Deviation); unit: months] | 59.36 (64.753) | 58.35 (61.834) | 58.85 (63.185)

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure on or After Week 2
Description: Treatment failure was defined by the occurrence of a uveitis flare (the inability to maintain disease control). To be considered treatment failure, ≥ 1 of these criteria had to be present in at least 1 eye at Week 2 or all other visits:
  * New active, inflammatory chorioretinal, and/or inflammatory retinal vascular lesions relative to Baseline
  * 2-step increase relative to Baseline in anterior chamber cell grade or vitreous haze grade
  * Worsening of best corrected visual acuity by ≥ 15 letters relative to baseline.
  Time to treatment failure was analyzed using the Kaplan-Meier method. Dropouts for reasons other than treatment failure at any time during the study were censored at the drop out date.
  Per protocol, the primary analysis was performed in the Main Study population which included all randomized participants recruited outside Japan; for completeness results are also reported below for the Integrated dataset which includes participants recruited in Japan.
Time Frame: From Baseline until end of study (up to 80 weeks)
Population: The intent-to-treat (ITT) population which included all randomized participants; 3 participants at 2 sites were excluded from the ITT due to incomplete efficacy source data and compliance issues.
Measure: Median (Inter-Quartile Range); unit: months
Groups:
- Main Study: Placebo: Participants, excluding those enrolled in the Japan sub-study, received placebo subcutaneous injection at Baseline followed by eow dosing starting at Week 1 for up to 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 10 - 35 mg/day at study entry followed by a protocol-defined mandatory taper until Week 19.
- Main Study: Adalimumab: Participants, excluding those enrolled in the Japan sub-study, received adalimumab 80 mg subcutaneous loading dose at Baseline followed by 40 mg doses eow starting at Week 1 for a maximum of 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 10 - 35 mg/day at study entry followed by a protocol-defined mandatory taper until Week 19.
- Integrated Study (Main + Japan Sub-study): Placebo: Participants, including those enrolled in the Main Study and the Japan Sub-study, received placebo subcutaneous injection at Baseline followed by eow dosing starting at Week 1 for up to 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 10 - 35 mg/day at study entry followed by a protocol-defined mandatory taper until Week 19.
- Integrated Study (Main + Japan Sub-study): Adalimumab: Participants, including those enrolled in the Main Study and the Japan Sub-study, received adalimumab 80 mg subcutaneous loading dose at Baseline followed by 40 mg doses eow starting at Week 1 for a maximum of 80 weeks or until treatment failure. Participants continued to receive prednisone orally, 10 - 35 mg/day at study entry followed by a protocol-defined mandatory taper until Week 19.
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 111 | 115 | 127 | 131
months | 8.3 [3.0 to NA] — Not estimable due to the low number of events | NA [4.7 to NA] — Not estimable due to the low number of events | 5.6 [2.6 to NA] — Not estimable due to the low number of events | NA [3.9 to NA] — Not estimable due to the low number of events
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; The primary analysis of the primary endpoint was performed on Main Study data, excluding the Japanese sub-study. The statistical test was performed at a 2-sided significance level of 0.05. The hazard ratio of adalimumab versus placebo was calculated using proportional hazards regression with treatment as factor; Test type: Superiority or Other; p = 0.004, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.39 to 0.84]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; An additional analysis of the primary endpoint was performed using the Integrated Study data (Main Study + Japan sub-study). The statistical test was performed at a 2-sided significance level of 0.05. The hazard ratio of adalimumab versus placebo was calculated using proportional hazards regression with treatment and race (Japanese versus non-Japanese) as factors; Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.37 to 0.74]

2. Secondary Outcome: Change in Anterior Chamber (AC) Cell Grade in Each Eye From Baseline to the Final/Early Termination Visit
Description: Slit lamp examinations were conducted at each visit to assess AC cell count. The number of AC cells observed within a 1 mm × 1 mm slit beam was used to determine the grade according to the Standardization of Uveitis Nomenclature (SUN) criteria:
  Grade 0 = < 1 cell
  Grade 0.5+ = 1 - 5 cells
  Grade 1+ = 6 - 15 cells
  Grade 2+ = 16 - 25 cells
  Grade 3+ = 26 - 50 cells
  Grade 4+ = > 50 cells.
Time Frame: Baseline and at the Final/Early Termination Visit (up to 80 weeks)
Population: Intent-to-treat population with a Baseline and at least one post-baseline value; last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 110 | 115 | 126 | 131
units on a scale
  Left eye | 0.57 (1.001) | 0.41 (0.969) | 0.61 (1.005) | 0.46 (0.996)
  Right eye | 0.53 (0.963) | 0.40 (0.927) | 0.60 (0.992) | 0.44 (0.950)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; The statistical test for the ranked secondary variables was carried out in hierarchical order at the significance level of 5%; Test type: Superiority or Other; p = 0.218, ANOVA; From ANOVA with treatment as factor adjusted for clustered observations (i.e., observations from each of the participant's eyes); Mean Difference = -0.14, 95% CI 2-sided [-0.37 to 0.08] — The mean difference between treatment groups with its 95% confidence interval is based on individual data from all eyes adjusted for correlated measurements within a subject in an analysis of variance (ANOVA) model
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.164, ANOVA; From ANOVA with treatment and race (Japanese versus non-Japanese) as factors adjusted for clustered observations; Mean Difference = -0.15, 95% CI 2-sided [-0.36 to 0.06] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Change in Vitreous Haze (VH) Grade in Each Eye From Baseline to the Final/Early Termination Visit
Description: Vitreous haze was measured using dilated indirect ophthalmoscopy (DIO) and assessed by the Investigator according to National Eye Institute (NEI) and SUN criteria:
  Grade 0: No evident vitreous haze;
  Grade 0.5+: Slight blurring of the optic disc margin because of the haze; normal striations and reflex of the nerve fiber layer cannot be visualized;
  Grade 1+: Permits a better definition of both the optic nerve head and the retinal vessels (compared to higher grades);
  Grade 2+: Permits better visualization of the retinal vessels (compared to higher grades);
  Grade 3+: Permits the observer to see the optic nerve head, but the borders are quite blurry;
  Grade 4+: Optic nerve head is obscured.
Time Frame: Baseline and Final/Early Termination Visit (up to 80 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 110 | 115 | 126 | 131
units on a scale
  Left eye | 0.33 (0.733) | 0.16 (0.601) | 0.35 (0.749) | 0.18 (0.614)
  Right eye | 0.27 (0.605) | 0.18 (0.604) | 0.36 (0.729) | 0.18 (0.602)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.070, ANOVA; From ANOVA of change from baseline to final/early termination visit with treatment as factor; Mean Difference = -0.13, 95% CI 2-sided [-0.28 to 0.01] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.016, ANOVA; From ANOVA with treatment and race (Japanese versus non-Japanese) as factors adjusted for clustered observations; Mean Difference = -0.17, 95% CI 2-sided [-0.31 to -0.03] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change In Logarithm of the Minimum Angle of Resolution (LogMAR) Best Corrected Visual Acuity (BCVA) In Each Eye From Baseline to the Final/Early Termination Visit
Description: Using corrective lenses based on that visit's refraction testing, participant's best corrected visual acuity was measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR chart. On the logMAR scale, 0 is equivalent to 20/20 visual acuity, the range of normal vision is considered to be from -0.2 - 0.1; higher values indicate visual impairment.
Time Frame: Baseline and Final/Early Termination Visit (up to 80 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 110 | 115 | 126 | 131
logMAR
  Left eye | 0.06 (0.239) | 0.01 (0.251) | 0.07 (0.230) | 0.02 (0.241)
  Right eye | 0.02 (0.198) | -0.01 (0.165) | 0.04 (0.216) | 0.00 (0.169)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.096, ANOVA; From ANOVA of change from baseline to final/early termination visit with treatment as factor adjusted for clustered observations; Mean Difference = -0.04, 95% CI 2-sided [-0.08 to 0.01] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.044, ANOVA; From ANOVA with treatment and race (Japanese versus non-Japanese) as factors adjusted for clustered observations; Mean Difference = -0.04, 95% CI 2-sided [-0.09 to 0.00] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Time to Optimal Coherence Tomography (OCT) Evidence of Macular Edema in At Least 1 Eye On or After Week 2
Description: Optical coherence tomography was performed at every visit using 1 of 3 approved machines. Images were evaluated by a central reader. Macular edema was defined as cystoid macular edema.
  OCT evidence of macular edema on or after Week 2 was to be counted as an event. Dropouts due to reasons other than OCT evidence of macular edema were to be considered as censored observations at the time of dropping out.
Time Frame: From Baseline until the Final Visit (up to 80 weeks)
Population: Intent to treat population with no macular edema at Baseline
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 95 | 90 | 106 | 102
months | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.491, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.34 to 1.69] — The hazard ratio of adalimumab versus placebo was calculated using proportional hazards regression with treatment as factor
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.185, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.28 to 1.28] — The hazard ratio of adalimumab versus placebo was calculated using proportional hazards regression with treatment and race (Japanese versus non-Japanese) as factors

6. Secondary Outcome: Percent Change in Central Retinal Thickness in Each Eye From Baseline to the Final/Early Termination Visit.
Description: Central retinal thickness was measured using OCT and assessed by a central reader.
Time Frame: Baseline and Final/Early Termination Visit (up to 80 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 108 | 114 | 124 | 130
percent change
  Left eye (N = 107, 114, 122, 130) | 6.4 (20.67) | 4.5 (29.82) | 6.3 (19.75) | 5.2 (29.91)
  Right eye (N = 108, 113, 124, 129) | 7.7 (28.88) | 5.4 (34.83) | 9.9 (30.79) | 3.9 (33.34)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.451, ANOVA; From ANOVA of change from baseline to final/early termination visit with treatment and OCT machine as factors adjusted for clustered observations; Mean Difference = -2.3, 95% CI 2-sided [-8.5 to 3.8] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.174, ANOVA; From ANOVA with treatment, race (Japanese versus non-Japanese) and OCT machine as factors adjusted for clustered observations; Mean Difference = -3.9, 95% CI 2-sided [-9.7 to 1.8] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Change in Visual Functioning Questionnaire 25 (VFQ-25) Total Score From Baseline to the Final/Early Termination Visit
Description: The National Eye Institute VFQ-25 is an ocular disease-specific survey that measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning, in addition to task-oriented domains related to daily visual functioning.
  The VFQ-25 consists of a base set of 25 vision-targeted questions plus an additional single-item general health rating question. The overall composite score ranges from 0 to 100, where higher scores or increases in score indicate better vision-related functioning.
Time Frame: Baseline and Final/Early Termination Visit (up 80 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 109 | 115 | 125 | 131
units on a scale | 1.24 (10.698) | 3.36 (11.73) | 1.00 (10.225) | 2.79 (12.018)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.160, ANOVA; From ANOVA of change from baseline to final/early termination visit with treatment as a factor; Mean Difference = 2.12, 95% CI 2-sided [-0.84 to 5.08]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.205, ANOVA; From ANOVA of change from baseline to final/early termination visit with treatment and race (Japanese versus non-Japanese) as factors; Mean Difference = 1.77, 95% CI 2-sided [-0.97 to 4.52]

8. Secondary Outcome: Change in VFQ-25 Subscore Distance Vision From Baseline to the Final/Early Termination Visit
Description: The National Eye Institute VFQ-25 is an ocular disease-specific survey that measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning, in addition to task-oriented domains related to daily visual functioning.
  The VFQ-25 consists of a base set of 25 vision-targeted questions plus an additional single-item general health rating question. The distance vision subscore is calculated from the answers to 3 distance vision-related questions and ranges from 0 to 100, where higher scores or increases in score indicate better vision-related functioning.
Time Frame: Baseline and Final/Early Termination Visit (up 80 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 109 | 115 | 125 | 131
units on a scale | 0.76 (16.248) | 2.64 (17.165) | 0.60 (15.978) | 2.96 (17.121)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.401, ANOVA; From ANOVA of change from baseline to final/early termination visit with treatment as a factor; Mean Difference = 1.88, 95% CI 2-sided [-2.53 to 6.29]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.256, ANOVA; [statistical method as in outcome 7, analysis 2]; Mean Difference = 2.36, 95% CI 2-sided [-1.73 to 6.45]

9. Secondary Outcome: Change in VFQ-25 Subscore Near Vision From Baseline to the Final/Early Termination Visit
Description: The National Eye Institute VFQ-25 is an ocular disease-specific survey that measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning, in addition to task-oriented domains related to daily visual functioning.
  The VFQ-25 consists of a base set of 25 vision-targeted questions plus an additional single-item general health rating question. The near vision subscore is calculated from the answers to 3 near vision-related questions and ranges from 0 to 100, where higher scores or increases in score indicate better vision-related functioning.
Time Frame: Baseline and Final/Early Termination Visit (up 80 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 109 | 115 | 125 | 131
units on a scale | 3.98 (17.397) | 3.88 (18.302) | 3.73 (17.17) | 2.89 (50.503)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.967, ANOVA; From ANOVA of change from baseline to final/early termination visit with treatment as a factor; Mena Difference = -0.10, 95% CI 2-sided [-4.81 to 4.61]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.714, ANOVA; [statistical method as in outcome 7, analysis 2]; Mean Difference = -0.87, 95% CI 2-sided [-5.53 to 3.79]

10. Secondary Outcome: Change in VFQ-25 Subscore Ocular Pain From Baseline to the Final/Early Termination Visit
Description: The National Eye Institute VFQ-25 is an ocular disease-specific survey that measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning, in addition to task-oriented domains related to daily visual functioning.
  The VFQ-25 consists of a base set of 25 vision-targeted questions plus an additional single-item general health rating question. The ocular pain subscore is calculated form the answers to 2 eye pain questions and ranges from 0 to 100, where higher scores or increases in score indicate less pain.
Time Frame: Baseline and Final/Early Termination Visit (up 80 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Main Study: Placebo | Main Study: Adalimumab | Integrated Study (Main + Japan Sub-study): Placebo | Integrated Study (Main + Japan Sub-study): Adalimumab
Number analyzed (Participants) | 109 | 115 | 125 | 131
units on a scale | 2.87 (17.233) | 3.42 (21.32) | 2.60 (17.339) | 2.15 (21.689)
Statistical Analysis 1: Comparison: Main Study: Placebo vs Main Study: Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.830, ANOVA; From ANOVA of change from baseline to final/early termination visit with treatment as a factor; Mean Difference = 0.56, 95% CI 2-sided [-4.56 to 5.68]
Statistical Analysis 2: Comparison: Integrated Study (Main + Japan Sub-study): Placebo vs Integrated Study (Main + Japan Sub-study): Adalimumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.842, ANOVA; From ANOVA of change from baseline to final/early termination visit with treatment and race (Japanese vs. non-Japanese) as factors; Mean Difference = -0.49, 95% CI 2-sided [-5.32 to 4.34]

ADVERSE EVENTS:
Time Frame: From the first study drug administration until 70 days following the last study drug administration or until rollover into the extension study. Median duration of treatment was 147 days in the placebo arm and 245 days in the adalimumab arm.
Arm/Group | Placebo | Adalimumab
Serious Adverse Events (participants affected / at risk) | 10/130 | 8/131
Other Adverse Events (participants affected / at risk) | 78/130 | 88/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=130) | Adalimumab (N=131)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 1
BLINDNESS TRANSIENT (Eye disorders) | 0 | 1
CHOROIDAL NEOVASCULARISATION (Eye disorders) | 1 | 0
RETINAL DETACHMENT (Eye disorders) | 1 | 0
SUBRETINAL FLUID (Eye disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 1
MENINGITIS ASEPTIC (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1
PNEUMONIA LEGIONELLA (Infections and infestations) | 0 | 1
TONSILLITIS (Infections and infestations) | 1 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
LUNG ADENOCARCINOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
DYSARTHRIA (Nervous system disorders) | 0 | 1
STATUS MIGRAINOSUS (Nervous system disorders) | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 | 1
AORTIC DISSECTION (Vascular disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=130) | Adalimumab (N=131)
CYSTOID MACULAR OEDEMA (Eye disorders) | 7 | 7
DRY EYE (Eye disorders) | 8 | 5
EYE PAIN (Eye disorders) | 6 | 9
UVEITIS (Eye disorders) | 9 | 6
VISUAL ACUITY REDUCED (Eye disorders) | 10 | 6
DIARRHOEA (Gastrointestinal disorders) | 9 | 4
NAUSEA (Gastrointestinal disorders) | 9 | 4
FATIGUE (General disorders) | 9 | 14
INJECTION SITE PAIN (General disorders) | 9 | 8
PYREXIA (General disorders) | 8 | 6
INFLUENZA (Infections and infestations) | 7 | 3
NASOPHARYNGITIS (Infections and infestations) | 20 | 23
SINUSITIS (Infections and infestations) | 4 | 8
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 10
URINARY TRACT INFECTION (Infections and infestations) | 11 | 13
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 9
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 8
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 | 28
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 10
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 10
HEADACHE (Nervous system disorders) | 17 | 17
INSOMNIA (Psychiatric disorders) | 3 | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 11
HYPERTENSION (Vascular disorders) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.